CLINICAL TRIAL: NCT05422937
Title: Symptom Patterns and Life With Longer Term COVID-19 in Children and Young People (SPLaT-19 Cohort & Qualitative Study)
Acronym: SPLaT-19
Status: Completed | Type: Observational
Sponsor: Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: RG-0348-22
Record Dates: First submitted 2022-06-16; First posted 2022-06-21 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: COVID-19; Pediatric ALL
MeSH Terms: conditions — COVID-19; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and Young People aged 8-17: All CYP aged 8 years - 17 years & 11 months whether they have had acute COVID-19 or not. Exposure to COVID-19 will be defined as a self-reported positive Sars-CoV-2 PCR test OR a positive self-reported OR self-reported presumed COVID-19 illness. Participants must have a recorded mobile number in their GP record.

SUMMARY:
Introduction:

While there is a substantial body of knowledge about acute Covid-19 in children and young people (CYP), less is known about long-COVID, where symptoms continue beyond four weeks, particularly since the most recent wave of the Omicron variant and the UK childhood vaccination programme roll out. This study aims to provide a picture of longer-term effects of an acute Covid-19 infection in CYP and identify their needs.

Methods and analysis:

The study comprises an observational prospective cohort study and a linked qualitative study. The cohort study will identify CYP aged 8-17 years in the West Midlands of England and, irrespective of Covid-19 status, invite them to complete an online questionnaire at point of recruitment, and after 3, 6, 9 and 12 months. CYP who have experienced long-term effects of COVID-19 will be invited to interview and, those who are currently experiencing symptoms, will be invited to record their experiences in a diary. Adults working in professional or third sector/voluntary roles with CYP will be invited to take part in a focus group to explore the perceived impact of Long-COVID on the wider experience of CYP. Approximately 900 participants will be needed for the cohort study to ensure the sample size is suitable, with approximately 20 CYP invited to interview and approximately 8 professionals invited to a focus group. Descriptive statistics will be used to describe incidence rates of symptoms and symptom resolution trajectories, and comparisons made between exposed and non-exposed groups. Logistic regression models will be used to estimate associations between candidate predictors and development of Long-COVID at each follow-up point. Linear regression will be used to estimate associations between candidate predictors and poor outcome in terms of health-related quality of life, as described by the KIDSCREEN10. Qualitative data will be analysed thematically using the constant comparison method.

Ethics and dissemination:

Research Ethics Committee and Health Research Authority approvals will be sought. Information about where to seek support will be provided to participants to mitigate against risks of harm. Study findings will be presented at conferences and published in open access journals.

ELIGIBILITY:
Inclusion Criteria for Cohort:

• All CYP aged 8 years - 17 years & 11 months will be eligible for the study regardless of whether they have had acute COVID-19 or not. Exposure to COVID-19 will be defined as a self-reported positive Sars-CoV-2 PCR test OR a positive self-reported LFD OR self-reported presumed COVID-19 illness. Participants must have a recorded mobile number in their GP record.

Exclusion Criteria for Cohort:

• CYP aged 8-17 (inclusive) who have relevant dissent codes on their medical records, indicating that their records are not to be used for research. CYP who have declined consent for text messaging services will not be invited to the study. CYP younger than 8 years and older than 17 years and 11 months will not be invited to the study.

Inclusion Criteria for Interviews:

• Children and adolescents (n≈20) aged 8 to 17 years, with evidence of Long COVID, as identified through participation in SPLaT cohort and defined as symptoms persisting longer than 4 weeks following an acute episode of COVID-19.

Inclusion Criteria for Focus Group:

• Adults working with children and adolescents in roles including teaching, social work, and voluntary organisations, identified by our local networks (n≈8).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All CYP aged 8 years - 17 years & 11 months (inclusive), registered at a participating general practice, will be invited to participate, subject to the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Screening For and Promotion of Health-Related Quality of Life in Children and Adolescents - a European Public Health perspective (KIDSCREEN, specifically using the KIDSCREEN 10 tool) | 12 months
  Global health-related quality of life measure. Minimum value 1 and maximum value 5 per question. Higher values indicate better quality of life.

SECONDARY OUTCOMES:
Inventory of Long COVID symptoms | 12 months
  Based on the ISARIC-WHO COVID-19 Survey and NICE COVID rapid evidence review
Health service utilisation | 12 months
  Contacts with and attendances at GP surgery, A&E attendance, referrals to secondary care (including paediatric fatigue clinic), hospital admission, contact with counselling / mental health services
New medical conditions diagnosed since COVID | 12 months
  Any new medical conditions diagnosed since COVID (e.g. asthma, type 1 diabetes)
School absence and attainment | 12 months
  Days absent and difficulties completing school work

CONTACTS AND LOCATIONS:
Locations (1):
- Keele University, Newcastle-under-Lyme, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Any requests for access to the data from anyone outside of the research team (e.g. collaboration, joint publication, data sharing requests from publishers) will follow the Keele University's data sharing procedure.